CLINICAL TRIAL: NCT02014441
Title: A Phase 2, Multicenter, Single-arm Trial to Evaluate the Biodistribution and Shedding of Talimogene Laherparepvec in Subjects With Unresected, Stage IIIB to IVM1c Melanoma
Brief Title: Single-arm Trial to Evaluate the Biodistribution and Shedding of Talimogene Laherparepvec
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120324
Record Dates: First submitted 2013-11-22; First posted 2013-12-18 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Talimogene Laherparepvec (Experimental): Talimogene laherparepvec was administered by intralesional injection into injectable cutaneous, subcutaneous, and nodal lesions at an initial dose of 10⁶ plaque-forming units (PFU) per mL followed by a dose of 10⁸ PFU/mL 21 days after the initial dose and every 14 days thereafter.
  Participants were treated with talimogene laherparepvec until they achieved a complete response (CR), all injectable tumors had disappeared, clinically relevant (resulting in clinical deterioration or requiring change of therapy) disease progression per modified World Health Organization (WHO) response criteria beyond 6 months of therapy, or intolerance of study treatment, whichever occurred first.
  Interventions: Drug: Talimogene laherparepvec

INTERVENTIONS:
Drug: Talimogene laherparepvec — Talimogene laherparepvec will be administered by intralesion injection at an initial dose of up to 4.0 mL of 10^6 PFU/mL. The second and subsequent doses will will be up to 4.0 mL 10^8 PFU/mL. The second dose should be administered 21 days from the initial dose. All subsequent doses should be given every 14 days.
  Other Names: IMLYGIC®; OncoVEX^GM-CSF

SUMMARY:
The primary objective was to estimate the proportion of participants with detectable talimogene laherparepvec deoxyribonucleic acid (DNA) in the blood and urine at any time after administration of talimogene laherparepvec within the first 3 cycles.

ELIGIBILITY:
Key Inclusion Criteria:

Male or female age ≥ 18 years with histologically confirmed diagnosis of melanoma and unresected stage IIIB, IIIC, IVM1a, IVM1b, or IVM1c regardless of prior line of therapy. Subject is candidate for intralesional therapy administration into cutaneous, subcutaneous, or nodal disease and must also have measurable disease, serum lactate dehydrogenase ≤ 1.5 x upper limit of normal, and Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and adequate hematologic, hepatic, and renal organ function.

Key Exclusion Criteria:

Subject must not have clinically active cerebral metastases, greater than 3 visceral metastases (this does not include lung metastases or any nodal metastases associated with visceral organs) or any bone metastases melanoma, primary ocular or mucosal melanoma, history or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or symptomatic autoimmune disease, or evidence of immunosuppression for any reason. Subject known to have acute or chronic active hepatitis B or hepatitis C infection, or human immunodeficiency virus infection will also be excluded. Subject who has active herpetic skin lesions or prior complications of herpes simplex virus type 1 ( HSV-1) infection (eg, herpetic keratitis or encephalitis), and/or requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use will also be excuded. Subject must not have received previous treatment with talimogene laherparepvec.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2016-01-25 (Actual); Study Completion 2018-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (14):
- United States (11):
  - Research Site, Tampa, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Fridley, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, New Brunswick, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Germantown, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Salt Lake City, Utah
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Montreal, Quebec

REFERENCES:
- [Background] Andtbacka RHI, Amatruda T, Nemunaitis J, Zager JS, Walker J, Chesney JA, Liu K, Hsu CP, Pickett CA, Mehnert JM. Biodistribution, shedding, and transmissibility of the oncolytic virus talimogene laherparepvec in patients with melanoma. EBioMedicine. 2019 Sep;47:89-97. doi: 10.1016/j.ebiom.2019.07.066. Epub 2019 Aug 10. PMID 31409575
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 centers in the United States and Canada. The first participant was enrolled on 07 April 2014 and the last participant was enrolled on 07 December 2015.
Groups:
- Talimogene Laherparepvec: Talimogene laherparepvec was administered by intralesional injection into injectable cutaneous, subcutaneous, and nodal lesions at an initial dose of 10⁶ plaque-forming units (PFU) per mL followed by a dose of 10⁸ PFU/mL 21 days after the initial dose and every 14 days thereafter.
Period: Overall Study
Arm/Group | Talimogene Laherparepvec
Started | 61
Received Treatment | 60
Completed | 49
Not Completed | 12
Not completed — Withdrawal by Subject | 12

BASELINE CHARACTERISTICS:
Population: Safety analysis set (all participants who received at least 1 dose of talimogene laherparepvec)
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 60
Eastern Cooperative Oncology Group (ECOG) Performance [Count of Participants; unit: Participants] — Scale to assess a patient's disease status.
  * 0 = Fully active, able to carry on all pre-disease performance without restriction;
  * 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature;
  * 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours;
  * 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours;
  * 4 = Completely disabled, confined to bed or chair;
  * 5 = Dead.
  Participants
    0 (Fully active) | 45
    1 (Restrictive but ambulatory) | 15
Herpes Simplex Virus Type 1 (HSV-1) Status [Count of Participants; unit: Participants] — HSV-1 status at baseline was determined by HSV-1 iimmunoglobulin G (IgG).
  Participants
    Negative | 17
    Positive | 40
    Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Deoxyribonucleic Acid (DNA) During the First Three Cycles
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of participants with detectable talimogene laherparepvec DNA in blood or urine at any time during cycles 1 to 3 is reported. The first cycle was 21 days in length, and subsequent cycles were 14 days in length.
Time Frame: Cycles 1 and 2 on days 1 (pre-dose and 1, 4, and 8 hours post-dose), 2, 3, 8, and 15 (cycle 1 only), cycle 3 on day 1 (pre-dose) and day 8, and cycle 4 on day 1 (pre-dose).
Population: Participants who were enrolled, received at least 1 dose of talimogene laherparepvec, and had at least 1 postdose blood/urine sample collected.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Talimogene Laherparepvec: HSV-1 Negative: Participants who were seronegative at baseline for HSV-1.
- Talimogene Laherparepvec: HSV-1 Positive: Participants who were seropositive at baseline for HSV-1.
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 60 | 17 | 40
percentage of participants
  Blood | 98.3 [91.1 to 100.0] | 100.0 [80.5 to 100.0] | 97.5 [86.8 to 99.9]
  Urine | 31.7 [20.3 to 45.0] | 29.4 [10.3 to 56.0] | 35.0 [20.6 to 51.7]

2. Secondary Outcome: Percentage of Participants With Clearance of Talimogene Laherparepvec DNA From Blood
Description: A participant was defined as having cleared talimogene laherparepvec if a negative blood sample was obtained following a prior positive test and if there were no subsequent positive tests.
Time Frame: as for outcome 1
Population: Participants must have received at least 1 dose of talimogene laherparepvec, had at least 2 post-dose blood samples collected within the same dosing cycle with at least 1 positive talimogene laherparepvec DNA sample and at least 1 subsequent sample at any time during the cycle.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 59 | 17 | 39
percentage of participants
  Cycle 1: number analyzed (Participants) | 41 | 14 | 25
  Cycle 1 | 92.7 [80.1 to 98.5] | 78.6 [49.2 to 95.3] | 100.0 [86.3 to 100.0]
  Cycle 2: number analyzed (Participants) | 57 | 17 | 38
  Cycle 2 | 86.0 [74.2 to 93.7] | 64.7 [38.3 to 85.8] | 94.7 [82.3 to 99.4]
  Cycle 3: number analyzed (Participants) | 3 | 2 | 1
  Cycle 3 | 33.3 [0.8 to 90.6] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5]

3. Secondary Outcome: Percentage of Participants With Clearance of Talimogene Laherparepvec DNA From Urine
Description: A participant was defined as having cleared talimogene laherparepvec if a negative urine sample was obtained following a prior positive test and if there were no subsequent positive tests.
Time Frame: as for outcome 1
Population: Participants received at least 1 dose of talimogene laherparepvec, had at least 2 post-dose urine samples collected within the same dosing cycle with at least 1 positive talimogene laherparepvec DNA sample and at least 1 subsequent sample at any time during the cycle.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 18 | 4 | 14
percentage of participants
  Cycle 1: number analyzed (Participants) | 3 | 1 | 2
  Cycle 1 | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0]
  Cycle 2: number analyzed (Participants) | 14 | 3 | 11
  Cycle 2 | 92.9 [66.1 to 99.8] | 100.0 [29.2 to 100.0] | 90.9 [58.7 to 99.8]
  Cycle 3: number analyzed (Participants) | 2 | 0 | 2
  Cycle 3 | 100.0 [15.8 to 100.0] |  | 100.0 [15.8 to 100.0]

4. Secondary Outcome: Percentage of Samples With Detectable Talimogene Laherparepvec DNA on the Exterior of the Occlusive Dressing During the First Three Cycles
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of swab samples from the exterior of the occlusive dressing with detectable talimogene laherparepvec DNA at any time during cycles 1 to 3 is reported.
Time Frame: Cycle 1 on days 2, 3, 8, and 15, cycle 2 on days 1 (pre-dose), 2, 3, and 8, cycle 3 on day 1 (pre-dose) and day 8, and cycle 4 on day 1 (pre-dose).
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab collected from the exterior of the occlusive dressing.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 60 | 17 | 40
Number analyzed (samples) | 1085 | 289 | 741
percentage of samples | 19.5 | 17.6 | 19.6

5. Secondary Outcome: Percentage of Samples With Detectable Talimogene Laherparepvec Virus on the Exterior of the Occlusive Dressing During the First Three Cycles
Description: If the result of the qPCR testing was positive, then a 50% tissue culture infective dose (TCID50) assay was performed on the swab sample to measure viral infectivity. The percentage of swab samples from the exterior of the occlusive dressing with detectable talimogene laherparepvec virus at any time during cycles 1 to 3 is reported.
Time Frame: as for outcome 4
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab collected from the exterior of the occlusive dressing with a detectable qPCR result.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 48 | 13 | 33
Number analyzed (samples) | 211 | 51 | 144
percentage of samples | 0.0 | 0.0 | 0.0

6. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA on the Exterior of the Occlusive Dressing During the First Three Cycles
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of participants with detectable talimogene laherparepvec DNA on the exterior of the occlusive dressing at any time during cycles 1 to 3 is reported.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 60 | 17 | 40
percentage of participants | 80.0 | 76.5 | 82.5

7. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Virus on the Exterior of the Occlusive Dressing During the First Three Cycles
Description: If the result of the qPCR testing was positive, then a 50% tissue culture infective dose (TCID50) assay was performed on the swab sample to measure viral infectivity. The percentage of participants with detectable talimogene laherparepvec virus on the exterior of the occlusive dressing at any time during cycles 1 to 3 is reported.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 48 | 13 | 33
percentage of participants | 0.0 | 0.0 | 0.0

8. Secondary Outcome: Percentage of Samples From the Surface of Injected Lesions With Detectable Talimogene Laherparepvec DNA During the First Three Cycles
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of swab samples from the surface of injected lesions with detectable talimogene laherparepvec DNA at any time during cycles 1 to 3 is reported.
Time Frame: as for outcome 4
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one injected lesion swab collected.
Measure: Number; unit: percentage of samples
Units Other Than Participants: Samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 60 | 17 | 40
Number analyzed (Samples) | 1260 | 307 | 885
percentage of samples | 57.6 | 53.7 | 57.3

9. Secondary Outcome: Percentage of Samples From the Surface of Injected Lesions With Detectable Talimogene Laherparepvec Virus During the First Three Cycles
Description: If the result of the qPCR testing was positive, then a 50% tissue culture infective dose (TCID50) assay was performed on the swab sample to measure viral infectivity. The percentage of samples taken from the surface of injected lesions with detectable talimogene laherparepvec virus at any time during cycles 1 to 3 is reported.
Time Frame: as for outcome 4
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one injected lesion swab collected with a positive qPCR result.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 60 | 17 | 40
Number analyzed (samples) | 725 | 165 | 506
percentage of samples | 1.1 | 3.0 | 0.6

10. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA on the Surface of Injected Lesions During the First Three Cycles
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of participants with detectable talimogene laherparepvec DNA swabs taken from the surface of injected lesions at any time during cycles 1 to 3 is reported.
Time Frame: as for outcome 4
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 60 | 17 | 40
percentage of participants | 100.0 | 100.0 | 100.0

11. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Virus on the Surface of Injected Lesions During the First Three Cycles
Description: If the result of the qPCR testing was positive, then a 50% tissue culture infective dose (TCID50) assay was performed on the swab sample to measure viral infectivity. The percentage of participants with detectable talimogene laherparepvec virus on swabs taken from the surface of injected lesions at any time during cycles 1 to 3 is reported.
Time Frame: as for outcome 4
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 60 | 17 | 40
percentage of participants | 11.7 | 23.5 | 7.5

12. Secondary Outcome: Percentage of Samples From Oral Mucosa With Detectable Talimogene Laherparepvec DNA During Treatment
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of swab samples from oral mucosa with detectable talimogene laherparepvec DNA at any time during treatment is reported.
Time Frame: Cycle 1 on days 1 (pre-dose), 8, and 15, cycles 2 and 3 on days 1 (pre-dose), and 8, cycle 4 and subsequent cycles (up to 47) on day 1 (pre-dose), cycle 25 on day 1 (pre-dose) and day 8.
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one oral mucosa swab collected during treatment.
Measure: Number; unit: percentage of samples
Units Other Than Participants: Samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 60 | 17 | 40
Number analyzed (Samples) | 964 | 302 | 599
percentage of samples | 1.2 | 2.6 | 0.5

13. Secondary Outcome: Percentage of Samples From Oral Mucosa With Detectable Talimogene Laherparepvec Virus During Treatment
Description: If the result of the qPCR testing was positive, then a 50% tissue culture infective dose (TCID50) assay was performed on the swab sample to measure viral infectivity. The percentage of samples taken from oral mucosa with detectable talimogene laherparepvec virus at any time during treatment is reported.
Time Frame: as for outcome 12
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one oral mucosa swab collected during treatment with a positive qPCR result.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 8 | 4 | 3
Number analyzed (samples) | 12 | 8 | 3
percentage of samples | 0.0 | 0.0 | 0.0

14. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA in Oral Mucosa During Treatment
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of participants with detectable talimogene laherparepvec DNA on swabs taken from oral mucosa at any time during treatment is reported.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 60 | 17 | 40
percentage of participants | 13.3 | 23.5 | 7.5

15. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Virus in Oral Mucosa During Treatment
Description: If the result of the qPCR testing was positive, then a 50% tissue culture infective dose (TCID50) assay was performed on the swab sample to measure viral infectivity. The percentage of participants with detectable talimogene laherparepvec virus in swabs taken from oral mucosa at any time during treatment is reported.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 8 | 4 | 3
percentage of participants | 0.0 | 0.0 | 0.0

16. Secondary Outcome: Percentage of Samples From the Anogenital Area With Detectable Talimogene Laherparepvec DNA During Treatment
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of swab samples from the anogenital area with detectable talimogene laherparepvec DNA at any time during treatment is reported.
Time Frame: Cycle 1 on days 1 (pre-dose), 8, and 15, cycles 2 and 3 on days 1 (pre-dose), and 8, cycle 4 and subsequent cycles (up to 50) on day 1 (pre-dose), Cycle 25 on day 1 (pre-dose) and day 8.
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab from the anogenital area collected during treatment.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 26 | 7 | 17
Number analyzed (samples) | 448 | 123 | 244
percentage of samples | 1.6 | 0.0 | 2.9

17. Secondary Outcome: Percentage of Samples With Detectable Talimogene Laherparepvec Virus in Swabs From the Anogenital Area During Treatment
Description: If the result of the qPCR testing was positive, then a 50% tissue culture infective dose (TCID50) assay was performed on the swab sample to measure viral infectivity. The percentage of samples with detectable talimogene laherparepvec virus in swabs taken from the anogenital area at any time during treatment is reported.
Time Frame: as for outcome 16
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab from the anogenital area collected during treatment with a positive qPCR result.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 5 | 0 | 5
Number analyzed (samples) | 7 | 0 | 7
percentage of samples | 0.0 |  | 0.0

18. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA in Swabs From the Anogenital Area During Treatment
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of participants with detectable talimogene laherparepvec DNA in swabs from the anogenital area at any time during treatment is reported.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 26 | 7 | 17
percentage of participants | 19.2 | 0.0 | 29.4

19. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Virus in Swabs From the Anogenital Area During Treatment
Description: If the result of the qPCR testing was positive, then a 50% tissue culture infective dose (TCID50) assay was performed on the swab sample to measure viral infectivity. The percentage of participants with detectable talimogene laherparepvec virus in swabs taken from the anogenital area at any time during treatment is reported.
Time Frame: as for outcome 16
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 5 | 0 | 5
percentage of participants | 0.0 |  | 0.0

20. Secondary Outcome: Percentage of Samples From Oral Mucosa With Detectable Talimogene Laherparepvec DNA After the End of Treatment
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of swab samples from oral mucosa with detectable talimogene laherparepvec DNA after the end of treatment is reported.
Time Frame: From 30 to 60 days after the last dose of talimogene laherparepvec (the median [minimum, maximum] duration of treatment was 23 [3, 141] weeks).
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one oral mucosa swab collected after the end of treatment.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 52 | 16 | 35
Number analyzed (samples) | 981 | 284 | 667
percentage of samples | 0.0 | 0.0 | 0.0

21. Secondary Outcome: Percentage of Samples From Oral Mucosa With Detectable Talimogene Laherparepvec Virus After the End of Treatment
Description: If the result of the qPCR testing was positive, then a 50% tissue culture infective dose (TCID50) assay was performed on the swab sample to measure viral infectivity.
Time Frame: as for outcome 20
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one oral mucosa swab collected after the end of treatment with a positive qPCR result.
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 0 | 0 | 0
Number analyzed (samples) | 0 | 0 | 0

22. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA in Oral Mucosa After the End of Treatment
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of participants with detectable talimogene laherparepvec DNA in swabs taken from oral mucosa after the end of treatment is reported.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 52 | 16 | 35
percentage of participants | 0.0 | 0.0 | 0.0

23. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Virus in Oral Mucosa After the End of Treatment
Description: as for outcome 21
Time Frame: as for outcome 20
Population: as for outcome 21
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Percentage of Samples From the Anogenital Area With Detectable Talimogene Laherparepvec DNA After the End of Treatment
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of swab samples from the anogenital area with detectable talimogene laherparepvec DNA after the end of treatment is reported.
Time Frame: as for outcome 20
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab from the anogenital area collected after end of treatment.
Measure: Number; unit: percentage of samples
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 21 | 7 | 13
Number analyzed (samples) | 515 | 187 | 326
percentage of samples | 0.0 | 0.0 | 0.0

25. Secondary Outcome: Percentage of Samples From the Anogenital Area With Detectable Talimogene Laherparepvec Virus After the End of Treatment
Description: as for outcome 21
Time Frame: 30 toFrom 30 to 60 days after the last dose of talimogene laherparepvec (the median [minimum, maximum] duration of treatment was 23 [3, 141] weeks). 60 days after the last dose of talimogene laherparepvec.
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab from the anogenital area collected after the end of treatment with a positive qPCR result.
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 0 | 0 | 0
Number analyzed (samples) | 0 | 0 | 0

26. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec DNA in Swabs From the Anogenital Area After the End of Treatment
Description: Talimogene laherparepvec DNA was measured using a quantitative polymerase chain reaction (qPCR) method. The percentage of participants with detectable talimogene laherparepvec DNA in swabs from the anogenital area after the end of treatment is reported.
Time Frame: as for outcome 20
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab from the anogenital area collected after the end of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 21 | 7 | 13
percentage of participants | 0.0 | 0.0 | 0.0

27. Secondary Outcome: Percentage of Participants With Detectable Talimogene Laherparepvec Virus in Swabs From the Anogenital Area After the End of Treatment
Description: as for outcome 21
Time Frame: as for outcome 20
Population: as for outcome 25
Arm/Group | Talimogene Laherparepvec | Talimogene Laherparepvec: HSV-1 Negative | Talimogene Laherparepvec: HSV-1 Positive
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Number of Samples With Detectable Talimogene Laherparepvec in Lesions Suspected to be Herpetic in Origin
Description: Any lesion such as a cold sore or vesicle thought to be herpetic in origin was evaluated by the investigator and swabbed if HSV infection was suspected. Quantitative PCR was performed on the swab sample to evaluate whether talimogene laherparepvec DNA was detectable in the sample.
Time Frame: From first dose until 60 days after last dose of talimogene laherparepvec; The median actual follow-up time was 28.9 weeks (range: 4 to 151 weeks).
Population: Participants who were enrolled, received at least one dose of talimogene laherparepvec, and had at least one swab sample collected from lesions suspected to be herpetic in origin during the study.
Measure: Number; unit: samples
Units Other Than Participants: samples
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 19
Number analyzed (samples) | 37
samples | 4

29. Secondary Outcome: Best Overall Response
Description: Response was assessed according to modified World Health Organization (WHO) criteria using both clinical (cutaneous, subcutaneous, or nodal tumor measurement by caliper) and radiological imaging (computed tomography (CT), magnetic resonance imaging (MRI), or ultrasound of the chest, abdomen, and pelvis and all other sites of disease).
  Complete response: disappearance of all index and non-index lesions.
  Partial Response: ≥ 50% reduction in size of all index lesions and any new measurable lesions.
  Stable disease: Neither sufficient tumor shrinkage of index lesion to qualify for response nor sufficient tumor increase of index lesion to qualify for progressive disease, assessed a minimum interval of 77 days from the first dose of study drug.
  Progressive Disease: ≥ 25% increase in size of index lesions or appearance of one or more non-index lesions.
Time Frame: Tumor response was assessed at weeks 12 and 24 and then at least every 3 months up to the end of treatment; median duration of treatment was 23.1 weeks (range: 3 to 141 weeks).
Population: All participants who received at least 1 dose of talimogene laherparepvec.
Measure: Number; unit: participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 60
participants
  Complete Response | 9
  Partial Response | 12
  Stable Disease | 10
  Progressive Disease | 26
  Unevaluable | 1
  Not Done | 2

30. Secondary Outcome: Objective Response Rate
Description: Response was assessed according to modified World Health Organization (WHO) criteria using both clinical (cutaneous, subcutaneous, or nodal tumor measurement by caliper) and radiological imaging (computed tomography, magnetic resonance imaging or ultrasound of the chest, abdomen, and pelvis and all other sites of disease). Objective response rate is defined as the percentage of participants with either a complete response or partial response. Subsequent confirmation was not required.
  Complete response: disappearance of all index and non-index lesions.
  Partial Response: ≥ 50% reduction in size of all index lesions and any new measurable lesions.
Time Frame: as for outcome 29
Population: All participants who received at least 1 dose of talimogene laherparepvec.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 60
percentage of participants | 35.0 [23.1 to 48.4]

31. Secondary Outcome: Time to Response
Description: Time to response was defined as the interval from the first dose of talimogene laherparepvec to the first event of complete response or partial response per modified WHO criteria; participants who did not respond were censored at the last evaluable tumor assessment.
Time Frame: as for outcome 29
Population: All participants who received at least 1 dose of talimogene laherparepvec.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 60
months | 8.7 [5.3 to NA] — Could not be estimated due to the low number of events

32. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was calculated only for those participants with an objective response and defined as the longest interval from an initial objective response (complete response or partial response) to disease progression per the modified WHO criteria or death, whichever occurred earlier; otherwise, DOR was censored at the last evaluable tumor assessment for participants who did not die or progress.
Time Frame: as for outcome 29
Population: All participants who received at least 1 dose of talimogene laherparepvec and had an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 21
months | NA [NA to NA] — Could not be estimated due to the low number of events

33. Secondary Outcome: Durable Response Rate
Description: Response was assessed according to modified World Health Organization (WHO) criteria using both clinical (cutaneous, subcutaneous, or nodal tumor measurement by caliper) and radiological imaging (computed tomography, magnetic resonance imaging or ultrasound of the chest, abdomen, and pelvis and all other sites of disease). Durable response rate is defined as the percentage of participants with a complete response or partial response maintained continuously for at least 6 months (183 days).
  Complete response: disappearance of all index and non-index lesions.
  Partial Response:≥ 50% reduction in size of all index lesions and any new measurable lesions.
Time Frame: as for outcome 29
Population: All participants who received at least 1 dose of talimogene laherparepvec.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 60
percentage of participants | 5.0 [1.0 to 13.9]

34. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the interval from first dose of talimogene laherparepvec to death from any cause; participants still alive were censored at the last known alive date.
Time Frame: as for outcome 28
Population: All participants who received at least 1 dose of talimogene laherparepvec.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 60
months | NA [NA to NA] — Could not be estimated due to the low number of events

35. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The Common Terminology Criteria for Adverse Events version 3.0 was used to grade severity of adverse events, based on the following general guideline: Grade 1 = Mild AE Grade 2 = Moderate AE Grade 3 = Severe AE Grade 4 = Life-threatening or disabling AE Grade 5 = Death related to AE. A serious adverse event was defined as an adverse event that meets at least 1 of the following serious criteria:
  * fatal
  * life threatening
  * requires in-patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event
  Treatment-related adverse events (TRAEs) are defined as adverse events possibly caused by talimogene laherparepvec, as assessed by the investigator.
Time Frame: From the first administration of talimogene laherparepvec up to 30 days after the last administration of talimogene laherparepvec; median duration of treatment was 23.1 weeks (range: 3 to 141 weeks).
Population: All participants who received at least 1 dose of talimogene laherparepvec.
Measure: Count of Participants; unit: Participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 60
Participants
  Any adverse event | 60
  AE grade ≥ 2 | 42
  AE grade ≥ 3 | 12
  AE grade ≥ 4 | 1
  Serious adverse events | 13
  AE leading to study drug discontinuation | 5
  Fatal AE | 0
  Treatment-related adverse event | 57
  Treatment-related AE grade ≥ 2 | 33
  Treatment-related AE grade ≥ 3 | 6
  Treatment-related AE grade ≥ 4 | 1
  Serious treatment-related AE | 8
  TRAE leading to study drug discontinuation | 3
  Fatal treatment-related AE | 0

ADVERSE EVENTS:
Time Frame: From the first administration of talimogene laherparepvec up to 30 days after the last administration of talimogene laherparepvec; median duration of treatment was 23.1 weeks (range: 3 to 141 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Talimogene Laherparepvec
Serious Adverse Events (participants affected / at risk) | 13/60
Other Adverse Events (participants affected / at risk) | 58/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (N=60)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Body temperature increased (Investigations) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Influenza like illness (General disorders) | 1
Pyrexia (General disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (N=60)
Abdominal distension (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 15
Nasopharyngitis (Infections and infestations) | 7
Oral herpes (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 4
Body temperature increased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 27
Somnolence (Nervous system disorders) | 4
Depression (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Night sweats (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 12
Skin lesion (Skin and subcutaneous tissue disorders) | 4
Hypotension (Vascular disorders) | 7
Stomatitis (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 7
Chest pain (General disorders) | 3
Chills (General disorders) | 39
Fatigue (General disorders) | 34
Influenza like illness (General disorders) | 12
Injection site erythema (General disorders) | 3
Injection site pain (General disorders) | 15
Injection site rash (General disorders) | 3
Injection site reaction (General disorders) | 6
Malaise (General disorders) | 3
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 15
Pyrexia (General disorders) | 23
Cellulitis (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Hypoaesthesia (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.